CLINICAL TRIAL: NCT02998398
Title: Evaluation of the Switch From the Original Infliximab ( REMICADE®) to Its Biosimilar (INFLECTRA®) in Daily Practice at Cochin Hospital
Brief Title: Evaluation of the Switch From the Original Infliximab to Its Biosimilar in Daily Practice at Cochin Hospital
Acronym: SIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI-16-004; 2016-A02016-A00700-51 (Other: ANSM)
Record Dates: First submitted 2016-05-17; First posted 2016-12-20 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Crohn's Disease; Uveitis
Keywords: Biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Crohn Disease; Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Switch from REMICADE® to INFLECTRA® — Treatment with an infliximab biosimilar (i.e. INFLECTRA® ) for all patients which have been treated by REMICADE® for at least 4 months

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the switch from the original infliximab ( REMICADE®) to its biosimilar (INFLECTRA®) in all the patients at Cochin hospital receiving REMICADE® for either a rheumatic, gastro-enterologic or ophthalmic condition

DETAILED DESCRIPTION:
All patients managed in one of the departments of cochin Hospital who are receiving the original infliximab ( REMICADE®) from at least 4 months will be invited to continue to receive infliximab but using its biosimilar (INFLECTRA®)) at the same regimen (identical dose per infusion and interval between two infusions) than the previous one while receiving REMICADE®. The tolerability of the infusion will be recorded as well as the percentage of patients continuing INFLECTRA® after at least six months of its initiation.

Moreover, the infliximab serum level will be evaluated after the last infusion of REMICADE® and after the third infusion of INFLECTRA®. At the same time, anti-drug antibodies will be tested.

Finally for each of the underlying disease (e.g. rheumatoid arthritis, spondyloarthritis, Crohn's disease, uveitis,..), the maintenance of the efficacy of Infliximab will be evaluated according to the usual outcome measures of the activity of the disease

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 18 year old
* Patient treated with REMICADE® in Cochin hospital
* More than 3 perfusions of REMICADE® before the switch to INFLECTRA®

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed in one of the departments of cochin Hospital who are receiving the original infliximab ( REMICADE®) from at least 4 months
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients continuing INFLECTRA® | after the third infusion of INFLECTRA®, up to 24 weeks
  Evaluation of the percentage of patients continuing INFLECTRA® after its third infusion

SECONDARY OUTCOMES:
Infliximab serum level | after the third infusion of INFLECTRA®, up to 24 weeks
Percentage of patients with a flare of their disease | after the third infusion of INFLECTRA®, up to 24 weeks
  The flare will be assessed by usual physiological parameter of the disease
Percentage of patients with anti-drug antibodies assessed after the third infusion of INFLECTRA® | after the third infusion of INFLECTRA®, up to 24 weeks
Percentage of patients with anti drug antibodies assessed after the last infusion of REMICADE® | after the last infusion of REMICADE®, up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maxime DOUGADOS, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Avouac J, Molto A, Abitbol V, Etcheto A, Salcion A, Gutermann L, Klotz C, Elhai M, Cohen P, Soret PA, Morin F, Conort O, Chast F, Goulvestre C, Jeunne CL, Chaussade S, Kahan A, Roux C, Allanore Y, Dougados M. Systematic switch from innovator infliximab to biosimilar infliximab in inflammatory chronic diseases in daily clinical practice: The experience of Cochin University Hospital, Paris, France. Semin Arthritis Rheum. 2018 Apr;47(5):741-748. doi: 10.1016/j.semarthrit.2017.10.002. Epub 2017 Oct 5. PMID 29102156